CLINICAL TRIAL: NCT00158652
Title: Phase III Trial Comparing Conventional RT With Concomitant CT Versus Accelerated RT With Concomitant CT Versus Very Accelerated RT Alone in Patients With Head and Neck Squamous Cell Carcinoma
Brief Title: Accelerated Radiotherapy and Concomitant Chemo-radiotherapy in HNSCC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Groupe Oncologie Radiotherapie Tete et Cou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GORTEC 99-02
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2011-11

CONDITIONS: Oral Cancer; Oropharynx Cancer; Hypopharynx Cancer; Larynx Cancer
Keywords: Head and neck squamous cell carcinoma; Radiotherapy; Chemotherapy
MeSH Terms: conditions — Mouth Neoplasms; Oropharyngeal Neoplasms; Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Fluorouracil; Carboplatin

ARMS (3):
- 1 (Active Comparator)
  Interventions: Procedure: Conventional radiotherapy 70 Gy in 7 weeks; Drug: 5FU, Paraplatin
- 2 (Experimental)
  Interventions: Procedure: middle accelerated radiotherapy 70 Gy in 6 weeks; Drug: 5FU, Paraplatin
- 3 (Experimental)
  Interventions: Procedure: very accelerated radiotherapy 64.8 Gy in 3.5 weeks

INTERVENTIONS:
Procedure: Conventional radiotherapy 70 Gy in 7 weeks — 2 gy per fraction, 1 fraction per day, 5 fractions per week
  Arms: 1
Procedure: middle accelerated radiotherapy 70 Gy in 6 weeks — 5 x 2gy/week until 40 Gy in 20 fractions and 4 weeks, then 2 fractions of 1.5Gy per day for 30 additional Gy in 2 weeks
  Arms: 2
Procedure: very accelerated radiotherapy 64.8 Gy in 3.5 weeks — 2 fractions of 1.8 Gy per day for 64.8 Gy in 3.5 weeks
  Arms: 3
Drug: 5FU, Paraplatin — 5FU 600mg/m²/D, Paraplatin 70mg/m²/D In arm 1: D1-4, 3 cycles during Rth (D1, D22, D43) In arm 2: D1-5, 2 cycles during Rth (D1, D29)
  Arms: 1; 2

SUMMARY:
This is a multicentric randomized phase III trial comparing conventional radiotherapy with concomitant chemotherapy versus accelerated radiotherapy with concomitant chemotherapy versus very accelerated radiotherapy in patients with stage III-IV head and neck squamous cell carcinoma. The main end point is the event free survival.

DETAILED DESCRIPTION:
This is a multicentric randomized phase III trial comparing conventional radiotherapy with concomitant chemotherapy (arm A) versus middle accelerated radiotherapy with concomitant chemotherapy (arm B) versus very accelerated radiotherapy alone (arm C) in patients with stage III-IV head and neck squamous cell carcinoma (HNSCC). The main end point is the event free survival.

The treatments are

Bras A : Conventional radiotherapy given once daily, delivering 70 Gy in 7 weeks (5 fractions of 2 Gy per week) and chemotherapy: 5FU : 600 mg/m²/d, Paraplatin : 70 mg/m²/d, D1-4 and D22-25 and D43-46

Bras B: middle accelerated radiotherapy delivering 70 Gy in 6 weeks and chemotherapy: 5FU : 600 mg/m²/d, Paraplatin : 70 mg/m²/d, D1-5 and D29-33

* first part : radiotherapy given once daily delivering 40 Gy in 4 weeks and 20 fractions of 2 Gy
* second part : radiotherapy given twice daily with "concomitant boost" delivering 30 Gy in 20 fractions in 2 weeks (1,5 Gy x 2 / day)

Bras C: very accelerated radiotherapy given twice daily delivering 64.8 Gy in 3.5 weeks in 36 fractions of 1.8 Gy

ELIGIBILITY:
Inclusion Criteria:

* Squamous cell carcinoma of oral cavity, oropharynx, hypopharynx or larynx
* Stage III-IV (UICC 1997): T2, T3 or T4 with N0-N3 or T0 with N2-N3
* Not resectable
* Karnofsky PS >= 70
* Renal/liver/cardiac functions and blood counts compatible with the use of paraplatin and 5-FU
* Informed consent signed

Exclusion Criteria:

* Distant metastasis
* Contra-indication to concomitant chemotherapy
* History of cancer
* History of head and neck radiotherapy

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 840 (Actual)
Dates: Start 2000-03; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Event free survival (event=progression, relapse, death from any cause) | 3 years

SECONDARY OUTCOMES:
Survival | 3 years
Loco regional control | 3 years
Toxicity | early and late

CONTACTS AND LOCATIONS:
Overall Officials: Jean Bourhis, PhD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris; Gilles Calais, Principal Investigator — CHU Tours
Locations (2):
- France (2):
  - CHU de Tours, Tours
  - Institut Gustave Roussy, Villejuif